CLINICAL TRIAL: NCT01791465
Title: Pilot Study of Extended-release Exenatide to Improve Glucose Control and Reduce Systemic Inflammation in Diabetic, HIV-infected Adults on Antiretroviral Therapy
Brief Title: Pilot Study of Bydureon to Treat Diabetes in HIV-infected Adults
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was terminated after 6 patients due to loss of funding
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, John R. Koethe, Assistant Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 121342; P30AI054999 (NIH)
Record Dates: First submitted 2013-02-11; First posted 2013-02-15 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Human Immunodeficiency Virus Infection; Diabetes Mellitus
Keywords: HIV; Diabetes
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bydureon treatment (Experimental): Treatment for 16 weeks with extended-release Exenatide (Bydureon)
  Interventions: Drug: extended-release exenatide

INTERVENTIONS:
Drug: extended-release exenatide — Single arm study - 2mg Bydureon every 7 days x 16 weeks
  Other Names: Bydureon

SUMMARY:
This pilot study will evaluate the effects of the anti-diabetic drug Bydureon (exenatide extended-release formulation) on blood sugar levels and serum markers of inflammation in a cohort of 12 HIV-infected adults on combination antiretroviral therapy (cART) with untreated diabetes mellitus. Previous studies have shown that high levels of persistent systemic inflammation predict the development of cardiovascular and metabolic diseases in HIV-infected persons on cART (a group at very high risk of atherosclerosis and myocardial infarction). Bydureon has demonstrated potent anti-inflammatory effects in prior studies of non-HIV infected persons, which suggests that this agent may represent a unique and preferred medication for the treatment of insulin resistance in HIV-infected adults. The Investigators hypothesize that short-term (16 weeks) therapy with Bydureon will improve glucose tolerance and significantly reduce circulating plasma levels of interleukin-6 (IL-6) and highly-sensitive C-reactive protein (hsCRP), two biomarkers strongly implicated in the development of cardiovascular and metabolic diseases in diabetic, HIV-infected, cART-treated adults.

DETAILED DESCRIPTION:
No further information. This was a single-arm trial to add an additional anti-diabetic medication to patients already known to be diabetic. The primary endpoint assessed whether the intervention reduced inflammation. There was no control arm.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Body mass index ≥ 25 kg/m2
* Glycosylated hemoglobin (A1C) value ≥ 6.5% OR having a fasting blood glucose ≥ 126 mg/dL
* On stable antiretroviral therapy for ≥ 12 months (with a fully suppressed plasma HIV-1 RNA level)
* Negative serum pregnancy test (females only)

Exclusion Criteria:

* History of pancreatitis
* Screening serum lipase value greater than or equal to 2 times the upper limit of normal (≥ 420 U/L)
* History of pancreatic cancer or thyroid cancer in patient, a first-degree relative, or a grandparent
* History of Multiple Endocrine Neoplasia (MEN) 2 syndrome
* History of gastroparesis, inflammatory bowel disease, and/or other severe gastrointestinal disease
* Estimated glomerular filtration rate (eGFR) ≤ 50 mls/minute
* Documented history of hypoglycemia (blood glucose <40 mg/dl)
* Active moderate-heavy alcohol use (more than 2 drinks/day) or >4 drinks in a single 24 hour period
* On an anti-diabetic medication within 3 months of enrollment
* On an HMG-CoA reductase inhibitor (statin) within 3 months of enrollment
* Persons on a didanosine (ddI) and/or stavudine (d4T)-containing cART (due to the heightened risk of pancreatitis)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Koethe, MD, Principal Investigator — Vanderbilt University School of Medicine; C. William Wester, MD, Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data is protected by HIPPA and Vanderbilt University research regulations. Summary de-identified data is available if requested

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Six HIV-infected participants recruited from the Vanderbilt Comprehensive Care Clinic between April 17, 2013 and May 6, 2016.
Pre-assignment Details: No consented participants were excluded prior to group assignment
Groups:
- Bydureon Treatment: Treatment for 16 weeks with extended-release Exenatide (Bydureon) extended-release exenatide. N=6 HIV-infected persons
Period: Overall Study
Arm/Group | Bydureon Treatment
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Bydureon Treatment: Treatment for 16 weeks with extended-release Exenatide (Bydureon) extended-release exenatide
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51 [45 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Serum Highly-sensitive C-reactive Protein (hsCRP) Levels at Baseline and 16 Weeks
Description: The primary outcome will be the change in hsCRP levels from baseline (pre-treatment) to 16 weeks of Bydureon treatment.
Time Frame: baseline and 16 weeks
Population: Change in hsCRP over 16 weeks of treatment
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
mg/dl
  baseline | 4.0 [2.0 to 14.9]
  16 weeks | 5.6 [2.4 to 20.3]
Statistical Analysis 1: Comparison: Bydureon Treatment; Test type: Superiority or Other; p = 0.08, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Serum Interleukin 6 (IL-6) at Levels at Baseline and 16 Weeks
Description: The primary outcome will be the change in serum IL-6 levels from baseline (pre-treatment) to 16 weeks of Bydureon treatment.
Time Frame: baseline and 16 weeks
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
mg/dl
  baseline | 1.07 [.68 to 3.01]
  week 16 | 1.27 [0.62 to 3.09]
Statistical Analysis 1: Comparison: Bydureon Treatment; The null hypothesis was that there would be no difference between baseline and 16 week IL-6; Test type: Superiority or Other; p = 0.34, Wilcoxon (Mann-Whitney) — Unadjusted - this was a Wilcoxon signed rank p-value (Baseline vs. week 16) comparison; no adjustments

3. Secondary Outcome: Serum Soluble Tumor Necrosis Factor Alpha (TNF-α) Levels at Baseline and 16 Weeks
Time Frame: baseline and 16 weeks
Measure: Mean (Inter-Quartile Range); unit: pg/ml
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
pg/ml
  baseline | 2.44 [1.73 to 3.74]
  16 weeks | 2.82 [2.4 to 3.90]
Statistical Analysis 1: Comparison: Bydureon Treatment; Test type: Superiority or Other; p = 0.046, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Serum Macrophage Chemotactic Protein-1 (MCP-1) Levels at Baseline and 16 Weeks
Time Frame: baseline and 16 weeks
Measure: Mean (Inter-Quartile Range); unit: pg/ml
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
pg/ml
  baseline | 5.73 [3.39 to 9.31]
  16 weeks | 4.78 [2.93 to 12.3]
Statistical Analysis 1: Comparison: Bydureon Treatment; Test type: Superiority or Other; p = 0.92, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Serum Macrophage Inflammatory Protein 1 Alpha (MIP-1 Alpha) Levels at Baseline and 16 Weeks
Time Frame: baseline and 16 weeks
Measure: Mean (Inter-Quartile Range); unit: pg/ml
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
pg/ml
  baseline | 0.088 [0.074 to 0.115]
  16 weeks | 0.081 [0.046 to 0.132]
Statistical Analysis 1: Comparison: Bydureon Treatment; Test type: Superiority or Other; p = 0.69, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Oral Glucose Insulin Sensitivity (OGIS) at Baseline and 16 Weeks
Description: The Oral Glucose Insulin Sensitivity (OGIS) is a method for the assessment of insulin sensitivity from the oral glucose tolerance test. OGIS provides an index which is analogous to the index of insulin sensitivity obtained from the glucose clamp. OGIS values for glucose clearance are reported in units of ml/min per square meter of body surface area. Lower values indicate slower glucose clearance and higher insulin resistance.
Time Frame: baseline and 16 weeks
Measure: Mean (Inter-Quartile Range); unit: ml/min/m^2 BSA
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
ml/min/m^2 BSA
  baseline | 310 [293 to 369]
  16 weeks | 399 [314 to 480]
Statistical Analysis 1: Comparison: Bydureon Treatment; Test type: Superiority or Other; p = 0.47, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Serum Adipokine Leptin Levels at Baseline and 16 Weeks
Time Frame: baseline and 16 weeks
Measure: Mean (Inter-Quartile Range); unit: ng/ml
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
ng/ml
  baseline | 17.4 [10.3 to 84.6]
  16 weeks | 14.3 [10.0 to 77.6]
Statistical Analysis 1: Comparison: Bydureon Treatment; Test type: Superiority or Other; p = 0.92, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Body Mass Index at Baseline and 16 Weeks
Time Frame: 16 weeks
Measure: Mean (Inter-Quartile Range); unit: kg/m2
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
kg/m2
  baseline | 32.6 [28.5 to 43.4]
  16 weeks | 31.3 [26.9 to 40.2]
Statistical Analysis 1: Comparison: Bydureon Treatment; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Serum TNF-a Receptor 1 Levels at Baseline and 16 Weeks
Time Frame: baseline and 16 weeks
Measure: Mean (Inter-Quartile Range); unit: pg/ml
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
pg/ml
  baseline | 392 [311 to 514]
  16 weeks | 399 [332 to 535]
Statistical Analysis 1: Comparison: Bydureon Treatment; Test type: Superiority or Other; p = 0.60, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Serum Soluble CD14 Levels at Baseline and 16 Weeks
Time Frame: baseline and 16 weeks
Measure: Mean (Inter-Quartile Range); unit: pg/ml
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
pg/ml
  baseline | 598 [458 to 802]
  16 weeks | 671 [562 to 805]
Statistical Analysis 1: Comparison: Bydureon Treatment; Test type: Superiority or Other; p = 0.08, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Serum TNF-a Receptor 2 Levels at Baseline and 16 Weeks
Time Frame: baseline and 16 weeks
Measure: Mean (Inter-Quartile Range); unit: pg/ml
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
pg/ml
  baseline | 598 [458 to 802]
  16 weeks | 671 [562 to 805]
Statistical Analysis 1: Comparison: Bydureon Treatment; Test type: Superiority or Other; p = 0.08, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Serum Hemoglobin A1c (HbA1c) Levels at Baseline and 16 Weeks
Time Frame: baseline and 16 weeks
Measure: Mean (Inter-Quartile Range); unit: percentage of glycated haemoglobin
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
percentage of glycated haemoglobin
  baseline | 7.6 [7.2 to 8.0]
  16 weeks | 6.3 [6.0 to 7.7]
Statistical Analysis 1: Comparison: Bydureon Treatment; Test type: Superiority or Other; p = 0.07, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Serum Triglycerides Levels at Baseline and 16 Weeks
Time Frame: baseline and 16 weeks
Measure: Mean (Inter-Quartile Range); unit: mg/dL
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
mg/dL
  baseline | 172 [100 to 245]
  16 weeks | 118 [110 to 189]
Statistical Analysis 1: Comparison: Bydureon Treatment; Test type: Superiority or Other; p = 0.69, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Serum Total Cholesterol Levels at Baseline and 16 Weeks
Time Frame: baseline and 16 weeks
Measure: Mean (Inter-Quartile Range); unit: mg/dL
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
mg/dL
  baseline | 192 [158 to 220]
  16 weeks | 176 [146 to 211]
Statistical Analysis 1: Comparison: Bydureon Treatment; Test type: Superiority or Other; p = 0.50, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Serum HDL Cholesterol Levels at Baseline and 16 Weeks
Time Frame: baseline and 16 weeks
Measure: Mean (Inter-Quartile Range); unit: mg/dL
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
mg/dL
  baseline | 39 [35 to 45]
  16 weeks | 34 [31 to 47]
Statistical Analysis 1: Comparison: Bydureon Treatment; Test type: Superiority or Other; p = 0.42, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Serum LDL Cholesterol Levels at Baseline and 16 Weeks
Time Frame: baseline and 16 weeks
Measure: Mean (Inter-Quartile Range); unit: mg/dL
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
mg/dL
  baseline | 127 [91 to 134]
  16 weeks | 109 [80 to 145]
Statistical Analysis 1: Comparison: Bydureon Treatment; Test type: Superiority or Other; p = 0.89, Wilcoxon (Mann-Whitney)

17. Other Pre Specified Outcome: Peripheral Endothelial Tonography, as Measured by the Non-invasive EndoPAT System Using the LnRHI (Natural Log of Reactive Hyperemia Index), at Baseline and 16 Weeks
Description: Normal: LnRHI > 0.51 Abnormal: LnRHI ≤ 0.51
Time Frame: baseline and 16 weeks
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
units on a scale
  baseline | 0.71 [0.42 to 0.93]
  16 weeks | 0.62 [0.59 to .77]
Statistical Analysis 1: Comparison: Bydureon Treatment; Test type: Superiority or Other; p = 0.75, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Body Weight at Baseline and 16 Weeks
Time Frame: baseline and 16 weeks
Measure: Mean (Inter-Quartile Range); unit: kilograms
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
kilograms
  baseline | 100 [87 to 112]
  16 weeks | 96 [81 to 111]
Statistical Analysis 1: Comparison: Bydureon Treatment; Test type: Superiority or Other; p = 0.046, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Waist Circumference at Baseline and 16 Weeks
Time Frame: baseline and 16 weeks
Measure: Mean (Inter-Quartile Range); unit: centimeters
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
centimeters
  baseline | 113 [105 to 134]
  16 weeks | 113 [102 to 132]
Statistical Analysis 1: Comparison: Bydureon Treatment; Test type: Superiority or Other; p = 0.25, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Hip Circumference at Baseline and 16 Weeks
Time Frame: baseline and 16 weeks
Measure: Mean (Inter-Quartile Range); unit: centimeters
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
centimeters
  baseline | 107 [102 to 125]
  16 weeks | 103 [97 to 117]
Statistical Analysis 1: Comparison: Bydureon Treatment; Test type: Superiority or Other; p = 0.12, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Waist to Hip Ratio at Baseline and 16 Weeks
Time Frame: baseline and 16 weeks
Measure: Mean (Inter-Quartile Range); unit: ratio
Arm/Group | Bydureon Treatment
Number analyzed (Participants) | 6
ratio
  baseline | 1.06 [1.03 to 1.07]
  16 weeks | 1.06 [1.05 to 1.12]
Statistical Analysis 1: Comparison: Bydureon Treatment; Test type: Superiority or Other; p = 0.046, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Bydureon Treatment
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bydureon Treatment (N=6)
Fatigue and weakness (General disorders) | 2 (2) — Self-reported

LIMITATIONS AND CAVEATS:
Trial terminated after only 6 individuals enrolled due to lack of interest in participation from patients and expiration of funding. Results are not considered reliable due to low number of observations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No